CLINICAL TRIAL: NCT06617429
Title: A Phase 3, Randomized, Double-blind, Sham-controlled Study Investigating the Efficacy and Safety of GTX-102 in Pediatric Subjects With Angelman Syndrome
Brief Title: Phase 3 Efficacy and Safety Study of GTX-102 in Pediatric Subjects With Angelman Syndrome (AS)
Acronym: Aspire
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTX-102-CL301; 2024-512600-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GTX-102 (Experimental): Participants will receive GTX-102 via lumbar puncture (LP) during both the double-blind and open-label period
  Interventions: Drug: GTX-102
- Sham-LP then GTX-102 (Sham Comparator): Participants will receive sham procedure during the double-blind period and then will receive GTX-102 via LP during the open-label period
  Interventions: Drug: GTX-102; Procedure: Sham-LP

INTERVENTIONS:
Drug: GTX-102 — antisense oligonucleotide
  Other Names: apazunersen
Procedure: Sham-LP — Small needle prick on the lower back at the location where the LP injection is normally made
  Arms: Sham-LP then GTX-102

SUMMARY:
The primary objective of this study is to evaluate the effect of GTX-102 in cognitive function in participants with deletion-type Angelman Syndrome (AS).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s)
* Confirmed diagnosis of AS with genetic confirmation of full maternal ubiquitin-protein ligase E3A (UBE3A) gene deletion causing AS in the region of 15q11.2 q13
* Able to ambulate independently, or with assistance at the Screening Visit (note, a child whose primary means of mobility is by wheelchair is excluded from the study)
* Platelet count, prothrombin time / international normalized ratio, and partial thromboplastin time within 1.5x the normal limits at the Screening Visit
* Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, and all study procedures, including LP procedure, MRI, and tolerating anesthesia without intubation
* From the time of informed consent through to at least 6 months after the final dose of GTX-102, females of childbearing potential who are sexually active must use highly effective contraception or abstinence. Males are able to participate if they agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the study and for at least 3 months after the final dose of GTX-102

Key Exclusion Criteria:

* Any change in medications or diet/supplements intended to treat symptoms of AS (eg, sleeping aids, antiseizure medications, supplements, dietary change including ketogenic or low-glycemic index diet, other) within the month prior to the Screening Visit (excluding weight-based adjustments)
* Any condition that creates an increased risk of unsuccessful LP
* Current or expected concomitant use of drugs that increase the risk of bleeding (eg, heparin, low molecular weight heparin, platelet inhibitors)
* Known hypersensitivity to GTX-102 or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
* Presence or history of any condition, lab abnormality, or infection, that, in the judgement of the Investigator, would interfere with participation, pose undue safety risk, or would confound interpretation of results
* Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 6 months or 5 half-lives prior to the Screening Visit or any prior use of gene therapy or ASO regardless of duration since last administration
* Concurrent participation in any interventional study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Bayley-4 Cognitive Raw Score Without Caregiver Input at Day 338 | Baseline, Day 338

SECONDARY OUTCOMES:
Net Response in Multidomain Responder Index (MDRI) | Day 338
Change from Baseline in ABC-C Hyperactivity/Noncompliance Subscale Score at Day 338 | Baseline, Day 338
Change from Baseline in Bayley-4 Receptive Communication Raw Score at Day 338 | Baseline, Day 338
Change from Baseline in Angelman Severity Assessment (ASA) Sleep Rating Raw Score at Day 338 | Baseline, Day 338
Change from Baseline in Vineland Adaptive Behavior Scales-3 (Vineland-3) Receptive Communication Raw Score at Day 338 | Baseline, Day 338
Change from Baseline in Vineland-3 Expressive Communication Raw Score at Day 338 | Baseline, Day 338
Change from Baseline in Bayley-4 Gross Motor Raw Score at Day 338 | Baseline, Day 338
Change from Baseline in ASA Gross Motor Rating at Day 338 | Baseline, Day 338
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), Severity of AEs and Relationship to Investigational Drug, Procedure, and Premedication | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc.
Locations (28):
- United States (14):
  - Cedars Sinai, Los Angeles, California
  - UCSD, Rady Children's Hospital, San Diego, California
  - UCSF, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - UNC Chapel Hill Pediatrics, Chapel Hill, North Carolina
  - Rare Disease Research, Hillsborough, North Carolina
  - The University of Texas, Austin, Texas
  - Carum Research Inc, Dallas, Texas
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - British Columbia Children's Hospital, Vancouver
- Germany (3):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - University of Leipzig, Leipzig
  - Haunersche Kinderklinik, Munich
- Japan (3):
  - Nagoya City University Graduate School of Medical Sciences, Nagoya, Aichi-ken
  - Osaka City General Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
- Poland (2):
  - Medical University of Gdańsk, Gdansk
  - Polish Mothers Memorial Institute, Lodz
- Spain (4):
  - Hospital Universitario Parc Tauli, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy Website — https://www.ultrarareadvocacy.com/conditions-we-study/angelman-syndrome-as/
- See also: Ultragenyx Angelman Syndrome (AS) Research Study Opportunity — https://www.ultraclinicaltrials.com/angelman-syndrome-as/
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/